CLINICAL TRIAL: NCT03669510
Title: Assessment of the Neurosensory Alteration With Computer Guided Inferior Alveolar Nerve Lateralization Versus Non Guided Classic Technique
Brief Title: Assessment of the Neurosensory Alteration After Inferior Alveolar Nerve Lateralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Reda Mohamed Abdelhady (Other)
Responsible Party: Sponsor-Investigator, Mohamed Reda Mohamed Abdelhady, director, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14422016552019
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Intervention Model Description: atrophic posterior mandible requiring nerve lateralization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer gaiuded IAN (Active Comparator): Computer guided surgical technique
  Interventions: Other: computer guided IAN lateralization surgical technique
- Classical technique (Experimental): Non computer guided surgical technique
  Interventions: Other: computer guided IAN lateralization surgical technique

INTERVENTIONS:
Other: computer guided IAN lateralization surgical technique — Tthe neurosensory alterations with computer guided inferior alveolar nerve lateralization versus non guided classic technique

SUMMARY:
: Assessment of the neurosensory alteration with computer guided inferior alveolar nerve lateralization versus non guided classic technique and measuring stability of implant after placement

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with with atrophied posterior mandibular ridge
* both sexes
* NO intra oral soft and hard tissue pathology
* NO systematic that contraindicate implant placement

Exclusion Criteria:

* Presence pathological lesion
* Heavy smokers more than 20 cigarettes per day.
* patients with systemic disease that may affect normal healing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the neurosensory alteration- sensation over time subjective(a scale 1-10) | 1 year
  assessing the sensation regaining over time subjective (a scale 1-10 )

SECONDARY OUTCOMES:
Implant stability | At the placement and after exposure ( up to 6 months )
  Measurements of the implant stability immediately after placement by osstell

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided